CLINICAL TRIAL: NCT03916211
Title: Clinical Study of Adipose-derived Stem Cells in the Treatment of Diabetic Foot
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maoquan Li (Other)
Responsible Party: Sponsor-Investigator, Maoquan Li, Prof. Dr. Li, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC-2018-04-02
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus Foot Ulcer
Keywords: stem cells
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine treatment (No Intervention): Diabetic foot routine treatment without intervention
- MSCs treatment (Experimental): On the basis of routine treatment of diabetic foot, adipose stem cells will be added to treat diabetic foot
  Interventions: Biological: MSCs treatment

INTERVENTIONS:
Biological: MSCs treatment — intramuscular injection of adipose stem cells treat diabetic foot
  Arms: MSCs treatment

SUMMARY:
1. Program Name: Clinical Study on Treatment of Diabetic Foot with Autologous Adipose Stem Cells
2. Bidding Unit: Tenth People's Hospital Affiliated to Tongji University
3. Study subjects: diabetic foot patients
4. OBJECTIVE: To establish an autologous adipose stem cell therapy for diabetic foot and evaluate its clinical safety and efficacy.
5. Study Design: Randomized Controlled Clinical Study
6. Target number of cases: 60
7. Main evaluation indicators: ulcer healing and amputation, calculating ulcer healing rate = total wound healing cases / total ulcer cases in this group; amputation rate = amputation cases / total cases in this group.
8. Secondary evaluation indicators: ankle-brachial index (ABI), Ruthford classification, painless walking time Wong-Baker Faces pain score, transcutaneous partial pressure of oxygen (TcPO2), laser Doppler flowmetry, multi-slice spiral CT angiography (CTA)

DETAILED DESCRIPTION:
research design: A randomized controlled trial was designed. According to the established inclusion criteria/exclusion criteria, the subjects were randomly divided into two groups by random number table. Each group received Mesenchymal Stem Cells(MSCs)from fat sources and conventional diabetic foot treatment according to the estimated results of sample size. A randomized controlled study was conducted with three blinds. The subjects were blind, the interventions were blind, and the evaluators were blind. Subjects were randomly grouped and assisted by coordinators. Follow-up was carried out at 5 time points 7 days, 1, 3, 6 and 12 months after operation to evaluate the pain and functional changes of the subjects, and to evaluate the safety and effectiveness.

Subject inclusion, exclusion criteria and allocation methods entry criteria and exclusion criteria will be executed.

Method of allocation and grouping:

A randomized controlled study was conducted with three blinds. The subjects were blind, the interventions were blind, and the evaluators were blind. Subjects were randomly grouped and assisted by coordinators. After receiving the random number, the test specimens and injections are marked by the research number rather than the names of the subjects. Injections of stem cells or saline are randomly determined by the computer system and will not be disclosed to the subjects. Subject groups would not inform the interveners that each injection was prepared by an assistant and the syringe was covered with black cloth. The operator and the participants would not know which drug was injected. The evaluation is done by a third party and the grouping will not be disclosed to the evaluator.After preliminary screening of qualified subjects, after signing the informed consent and verifying the entry/exclusion criteria by the research unit, and confirming that they meet the selection criteria, according to the results of the random system, the distribution of subjects is strictly carried out according to the random results.Subject Entry Records: Researchers should fill in the corresponding record forms according to the order of participants'enrollment, including the screening form, the identification form and the record form of participants' enrollment. All research-related test sheets need to be attached to the original record sheet kept by the researcher. The original record table is also the original record of this study which is monitored according to Good Clinical Practice(GCP)principle.

Number of cases required:

To test the effectiveness of stem cell therapy in the treatment of lower limb ischemic necrosis in diabetic patients, the subjects were randomly divided into stem cell treatment group and control group. Both groups received routine treatment, while the stem cell treatment group would receive stem cell therapy. According to the results of Lu Debin et al., the effective rate of stem cell therapy for ischemic necrosis of lower limbs in diabetic patients can reach 83.3%, while the effective rate in control group is 45%. In this study, two-sided test will be used, taking alpha = 0.05, beta = 0.1, and calculating the sample size according to the following formula .N=(Ualpha+Ubeta)22P(1-P)/(P1-P)2 N is the sample size required for each treatment group. In this study, the sample size was divided into two groups, and the sample size of each group was the same.

Ualpha and Ubeta are the standard normal deviations corresponding to alpha and beta respectively. Looking at the quantile table of normal distribution, we can see that Ualpha(0.05)=1.65, Ubeta(0.1)=1.28.

P 0 and P 1 represent the effective rates of the control group and the stem cell treatment group respectively. In this study, P 0 = 45%, P 1 = 83.3%; P = (P 0 + P 1) / 2 = (0.45 + 0.8333) / 2 = 0.6416, The above parameters and numerical values are introduced into the formula calculation.

N=(1.65+1.28)2*2*0.6416(1-0.6416)/(0.833-0.45)2=26.8732≈27 There were 54 patients in the two groups. Considering that some patients might withdraw from the study, the original sample size was added to 10% of the sample size, and the final sample size of the study was 60.

Use, dosage, time and course of treatment of stem cell preparations:

1. Stem cell preparation: stem cells derived from autologous fat.
2. Usage: Lower extremity muscle injection. Adipose stem cell transplantation anesthesia was performed by lumbar anesthesia; purified adipose stem cells were injected intramuscularly into lower extremities at intervals of 3 cm, which could be injected at about 50 points, 0.5 ml stem cell suspension at each point, about 1 x 106 cells, 25 points in lower extremities, 25 points in sole and well-being, and the total number of transplanted cells was about 1 x 108; (At the same time, the ulcer with infection was debrided and about 1 ml cell suspension was retained.) Subcutaneous injection of ulcer at the base and around the ulcer was performed, i.e. local injection of wound surface.
3. dose: The cells (1 x 108 cells) were mixed in 25 mL saline.
4. course of treatment: one-time intramuscular injection.

Criteria for discontinuation and termination of clinical research:

1. Research discontinuation 1.1 Subjects voluntarily withdraw from the study at any time without affecting further treatment.

   1.2 The following adverse events occurred (mainly referring to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) ).(1) fever, syncope, sweating, vomiting and other systemic symptoms with unknown causes; (2) dysfunction of gastrointestinal tract with unknown causes, loss of appetite, nausea, abdominal distention, constipation or diarrhea; (3) headache, fatigue, unexplained muscle pain, discomfort and changes in sleep; Mental symptoms such as anxiety, irritability, unexplained visual impairment, muscle tremor, dysuria, etc. Local manifestations such as skin macula, erythema, etc. Local pain aggravation or reduced range of activity, _Acute poisoning symptoms or death.

   1.3 Researchers believe that there are serious violations of research programs or incorrect grouping.

   1.4 Researchers believe that there are safety problems in the research program. 1.5 subjects were not interviewed. If participants discontinue treatment in advance, the cause of discontinuation must be documented in the Case report form (CRF), but follow-up is required until the end of the study and the study form is filled in.
2. Endpoint of the study 2.1 Severe treatment-related adverse events occurred between the end of treatment and the end of follow-up.

2.2 At the end of the follow-up, compared with the control group, ulcer healing, limb salvage rate, Ruthford grade, painless walking time, ankle-brachial index (ABI), transcutaneous partial pressure of oxygen (TcPO2), laboratory examination and vascular magnetic resonance imaging (MRA) improved significantly, indicating the effectiveness (with statistical differences): Criteria for evaluating efficacy

Compared with the control group, the ulcer healing rate, limb salvage rate, lower limb vascular ultrasound, ankle-brachial index (ABI), percutaneous partial pressure of oxygen (TcPO2), multi-slice spiral CT angiography (CTA), Rutherford grading, Wong-Baker Faces pain score of the subjects improved significantly compared with the control group, indicating the effectiveness (with statistical differences):

Main Evaluation Indicators:

1.Ulcer healing and amputation were calculated. Ulcer healing rate = number of complete wound healing cases / total number of ulcers in this group; amputation rate = number of amputations / total number of cases in this group.

2 Secondary Observation Indicators Lower extremity vascular ultrasound, ankle brachial index (ABI), percutaneous partial pressure of oxygen (TcPO2), multi-slice spiral CT angiography (CTA), Rutherford classification, Wong-Baker Faces pain score.

Recording requirements of adverse events and reporting methods and handling measures of serious adverse events Formulate detailed and standardized "Risk Management Mechanisms and Damage Event Processing Measures for Stem Cell Clinical Research" before the start of the experiment. All the subjects who received lower limb muscle injection of stem cells will become effective population for safety analysis. Researchers will faithfully record the side effects and adverse events of the subjects and analyze the causes.

1. Adverse events are defined as adverse and unexpected medical events during treatment and follow-up, including: (1) systemic symptoms such as fever, syncope, sweating and vomiting with unknown causes; (2) gastrointestinal dysfunction with unknown causes, anorexia, nausea, abdominal distention, constipation or diarrhea; and (3) headache, fatigue, unexplained muscle pain, No. Suitability and changes in sleep, etc. (4) Mental symptoms such as unexplained anxiety, restlessness and restlessness; (5) Visual impairment, muscle tremor, dysuria, etc. (5) Local manifestations such as skin macula and erythema; (5) Local pain aggravation or reduced range of activity; and (5) Acute poisoning symptoms or death.
2. Severe adverse events (SAEs) are defined as events requiring hospitalization, prolonging hospitalization, disability, impacting work ability, life-threatening or death-threatening, congenital malformations, etc. The severity of adverse events must be recorded and graded according to CTCAE criteria. The relationship between SAEs and treatment should be evaluated according to the following definitions. (1) Irrelevant: There is evidence that the cause of adverse events is not intra-articular injection therapy (such as past conditions, potential diseases, complications); 2) related: adverse events are time-related with intra-articular injection of drugs and known or suspected that intramuscular injection of drugs in lower extremities can cause the adverse events; 3) unable to assess. Adverse events are required to be recorded in the Case report form(CRF) related sections, which need to be described as: start and end dates; adverse event outcomes; whether they lead to withdrawal from the study; whether they are related to lower extremity intramuscular drug injections; and whether they are serious adverse events.

Reporting of Serious Adverse Events

Reporting time limit:

Within 24 hours of Observers'knowledge of the time of serious adverse events. Reporting mode Telephone or fax, and fill in the Record Form of Serious Adverse Events and send it to the main researchers, declaration units, ethics committees and the State Food and Drug Administration

ELIGIBILITY:
Inclusion Criteria:

* The age ranges from 30 to 65 years. There is no limit for male and female inpatients and outpatients who can be followed up.
* It conforms to the diagnostic criteria of diabetic foot of the sixth edition of Medical College Textbook Internal Medicine of the Ministry of Health.
* Severe lower limb ischemia (defined as resting ankle-brachial index (ABI) 0.4-0.8, accompanied by resting pain or intermittent claudication);
* The expected survival time is longer than one year.
* No human specific viruses (including HIV, HBV, HCV, HTLV, EBV, CMV, etc.) were detected and screened, and no Treponema pallidum infection was found.
* Voluntary subjects, the subjects understand the content of the experiment, and voluntarily sign the informed consent before the beginning of the experiment.

Exclusion Criteria:

* Diabetic retinopathy;
* There are allergies or contraindications to antiplatelet drugs, anticoagulants, thrombolytics, contrast agents, salicylates, etc.
* Haemorrhagic tendency, coagulation dysfunction, hypercoagulable constitution or refusal of transfusion therapy exist.
* In the past five years, patients with malignant diseases or markedly elevated levels of tumor markers in the blood were definitely diagnosed (the estimated survival time was less than 12 months).
* Pre-acute infectious disease symptoms;
* Patients with severe liver diseases (such as ascites, esophageal varices, liver transplantation, etc.); hemodynamic instability; renal failure undergoing dialysis; immunosuppressive therapy; decompensated heart failure (New York Heart Association Class III or IV) or myocardial infarction or bypass heart transplantation within three months before the start of the study; Hemorrhagic or ischemic stroke within 3 months before onset;
* Patients who are still participating in other clinical trials;
* Other researchers consider that patients who are not eligible for enrollment have other concomitant diseases.
* Subjects who refused to sign the informed consent or participate in the clinical trial.
* Immunodeficiency patients;

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-20 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
ulcer healing rate | up to 4 weeks
  Ulcer healing rate = number of cases of complete wound healing / total number of ulcers in this group
amputation rate | up to 4 weeks
  Amputation rate = number of amputations / total number of amputations in this group

SECONDARY OUTCOMES:
ultrasound | 2 weeks
  Evaluate patients' limbs blood flow by ultrasound，We will record blood flow velocities, for example， 4ml/second.
ABI(ankle brachial index) | 2weeks
  The ratio of ankle artery pressure to brachial artery pressure was obtained by measuring the contractile pressure of the posterior tibial artery, anterior tibial artery and brachial artery of the ankle.ABI≥0.9 means normal,0.8≥ABI≥0.7means mild arterial obstruction,0.6≥ABI≥0.4means moderate arterial obstruction,ABI<0.4means severe arterial obstruction.
TcPO2（Transcutaneous oxygen pressure） | 2 weeks
  Evaluate patients'oxygen level by TcPO2,TcPO2<20mmHg means very severe lesion.
CTA(Computed Tomography angiography) | up to 4 weeks
  Evaluate patients' limbs blood flow by CTA,We will record blood flow velocities, for example， 4ml/second.
Rutherford Classification | 2 weeks
  Evaluate patients' limbs blood flow by Rutherford classification，Grade 0: Normal Grade 1: Walking over 500 meters with lameness Grade 2: Walking 200-500 meters with lameness Grade 3: Walking within 200 meters with lameness Grade 4: Resting pain Grade 5: Small ulcer Grade 6: Large ulcer.
Wong-Baker Faces Pain Rating Scale | up to 4 weeks
  Evaluate patients' degree of pain by Wong-Baker Faces Pain Rating Scale.There are 6 faces in the Wong-Baker Pain Scale. The first face represents a pain score of 0, and indicates "no hurt". The second face represents a pain score of 2, and indicates "hurts a little bit." The third face represents a pain score of 4, and indicates "hurts a little more". The fourth face represents a pain score of 6, and indicates "hurts even more". The fifth face represents a pain score of 8, and indicates "hurts a whole lot"; the sixth face represents a pain score of 10, and indicates "hurts worst.

CONTACTS AND LOCATIONS:
Overall Officials: Li Xue, ph.D, Study Director — Shanghai 10th People'sHospital

REFERENCES:
- [Background] Lu Debin, Jiang Youzhao, Liang Ziwen, Li Xiaoyan, Zhang Zhonghui, Chen Bing.Autologous transplantation of bone marrow mesenchymal stem cells on diabetic patients with lower limb ischemia.Journal of Medical Colleges of PLA 2008;23:106-115
- [Background] Carlin JB, Doyle LW. Sample size. J Paediatr Child Health. 2002 Jun;38(3):300-4. doi: 10.1046/j.1440-1754.2002.00855.x. No abstract available. PMID 12047701
- [Background] Al-Delaimy WK, Merchant AT, Rimm EB, Willett WC, Stampfer MJ, Hu FB. Effect of type 2 diabetes and its duration on the risk of peripheral arterial disease among men. Am J Med. 2004 Feb 15;116(4):236-40. doi: 10.1016/j.amjmed.2003.09.038. PMID 14969651
- [Background] Khattab AD, Ali IS, Rawlings B. Peripheral arterial disease in diabetic patients selected from a primary care setting: Implications for nursing practice. J Vasc Nurs. 2005 Dec;23(4):139-48. doi: 10.1016/j.jvn.2005.09.005. PMID 16326332
- [Background] Rathur HM, Boulton AJ. The diabetic foot. Clin Dermatol. 2007 Jan-Feb;25(1):109-20. doi: 10.1016/j.clindermatol.2006.09.015. PMID 17276208
- [Background] Dick F, Diehm N, Galimanis A, Husmann M, Schmidli J, Baumgartner I. Surgical or endovascular revascularization in patients with critical limb ischemia: influence of diabetes mellitus on clinical outcome. J Vasc Surg. 2007 Apr;45(4):751-61. doi: 10.1016/j.jvs.2006.12.022. Epub 2007 Feb 15. PMID 17306950
- [Background] Engelhardt M, Bruijnen H, Scharmer C, Jezdinsky N, Wolfle K. Improvement of quality of life six months after infrageniculate bypass surgery: diabetic patients benefit less than non-diabetic patients. Eur J Vasc Endovasc Surg. 2006 Aug;32(2):182-7. doi: 10.1016/j.ejvs.2006.02.007. Epub 2006 Mar 29. PMID 16567116
- [Background] Huang P, Li S, Han M, Xiao Z, Yang R, Han ZC. Autologous transplantation of granulocyte colony-stimulating factor-mobilized peripheral blood mononuclear cells improves critical limb ischemia in diabetes. Diabetes Care. 2005 Sep;28(9):2155-60. doi: 10.2337/diacare.28.9.2155. PMID 16123483
- [Background] Humpert PM, Bartsch U, Konrade I, Hammes HP, Morcos M, Kasper M, Bierhaus A, Nawroth PP. Locally applied mononuclear bone marrow cells restore angiogenesis and promote wound healing in a type 2 diabetic patient. Exp Clin Endocrinol Diabetes. 2005 Oct;113(9):538-40. doi: 10.1055/s-2005-872886. PMID 16235157
- [Background] Canizo MC, Lozano F, Gonzalez-Porras JR, Barros M, Lopez-Holgado N, Briz E, Sanchez-Guijo FM. Peripheral endothelial progenitor cells (CD133 +) for therapeutic vasculogenesis in a patient with critical limb ischemia. One year follow-up. Cytotherapy. 2007;9(1):99-102. doi: 10.1080/14653240601034708. PMID 17354105
- [Background] Kern S, Eichler H, Stoeve J, Kluter H, Bieback K. Comparative analysis of mesenchymal stem cells from bone marrow, umbilical cord blood, or adipose tissue. Stem Cells. 2006 May;24(5):1294-301. doi: 10.1634/stemcells.2005-0342. Epub 2006 Jan 12. PMID 16410387
- [Background] De Ugarte DA, Morizono K, Elbarbary A, Alfonso Z, Zuk PA, Zhu M, Dragoo JL, Ashjian P, Thomas B, Benhaim P, Chen I, Fraser J, Hedrick MH. Comparison of multi-lineage cells from human adipose tissue and bone marrow. Cells Tissues Organs. 2003;174(3):101-9. doi: 10.1159/000071150. PMID 12835573
- [Background] Zuk PA, Zhu M, Ashjian P, De Ugarte DA, Huang JI, Mizuno H, Alfonso ZC, Fraser JK, Benhaim P, Hedrick MH. Human adipose tissue is a source of multipotent stem cells. Mol Biol Cell. 2002 Dec;13(12):4279-95. doi: 10.1091/mbc.e02-02-0105. PMID 12475952
- [Background] Gimble JM, Katz AJ, Bunnell BA. Adipose-derived stem cells for regenerative medicine. Circ Res. 2007 May 11;100(9):1249-60. doi: 10.1161/01.RES.0000265074.83288.09. PMID 17495232
- [Background] Wei Y, Hu H, Wang H, Wu Y, Deng L, Qi J. Cartilage regeneration of adipose-derived stem cells in a hybrid scaffold from fibrin-modified PLGA. Cell Transplant. 2009;18(2):159-70. doi: 10.3727/096368909788341261. PMID 19499704